CLINICAL TRIAL: NCT02258711
Title: SIgns and Symptoms Self-Monitoring and Psychoeducation in bipoLar Patients With a Smart-phonE Application (SIMPLE)
Brief Title: Self-Monitoring and Psychoeducation in Bipolar Patients With a Smart-phone Application
Acronym: SIMPLE
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical problems.
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); Institut Hospital del Mar d'Investigacions Mèdiques (IMIM) (Unknown); Centro de Investigación Biomédica en Red de Salud Mental (Network); Sodep S.A. (Unknown)
Responsible Party: Principal Investigator, Diego Hidalgo-Mazzei, Diego Hidalgo-Mazzei, M.D., Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCPPFR02062014
Record Dates: First submitted 2014-10-03; First posted 2014-10-07 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder; Psychoeducation; Smart-phone monitoring
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SIMPLe 2.0 plus Treatment as Usual (TAU) (Experimental): Psychoeducative and self-monitoring smart-phone application plus treatment as usual which includes pharmacological and psychological treatment.
  Interventions: Device: SIMPLE 2.0
- Treatment as usual (TAU) (No Intervention): Treatment as usual which includes pharmacological and psychological treatment.

INTERVENTIONS:
Device: SIMPLE 2.0 — SIMPLE 2.0 psychoeducative and self-monitoring smart-phone application plus treatment as usual.
  Arms: SIMPLe 2.0 plus Treatment as Usual (TAU)

SUMMARY:
Bipolar disorder is a frequent condition in the general population with a high morbimortality, which consists in dysfunctional temporal fluctuations between different mood phases ranging from depression to manic episodes with frequent subsyndromal symptoms between them. Usually during these phases, the subjects have a lack of insight about the diagnosis and symptoms. Besides the pharmacological treatment, additional psychological interventions have shown to improve the long-term outcome of the disorder, yet taking into account the limited resources currently available, its general implementation is still difficult and costly. Among these interventions, group psychoeducational programs have proved to be cost-effective in helping patients recognize early signs and symptoms in order to prevent full blown episodes which very usually are associated with a high morbidity and hospital admissions.

On the other hand, numerous projects have tested the potential benefits of new technologies such internet in the treatment of bipolar and psychotic disorders patients using either online signs and symptoms monitoring or web-based psychoeducational programs, yet to the investigators knowledge, none of them have integrated both approaches in one single intervention.

The hypothesis that, combining both interventions (signs and symptoms monitoring along with psychoeducational contents) in a single smart-phone application will prove to be at least equal or superior in terms of efficacy comparing to the standard treatment, seems promising, given the fact that both approaches have independently demonstrated their efficacy in the same population. This could extend the range of the patients in whom this kind of additional interventions could be implemented; preventing relapses, suicide attempts, consultations and hospitalizations at a much lower cost.

DETAILED DESCRIPTION:
The main aim of this study is to develop and clinically validate a smart-phone application to monitor symptoms and signs in stable bipolar patients, offering also customized embedded psycho-education contents and empower the self-management of their disorder to avoid relapses and hospitalizations. Secondary objectives will be to explore other clinical benefits among the smart-phone application users such as biological rhythms, manic/hypomanic and depressive symptoms, quality of life, suicide attempts, pharmacological treatment changes as well as healthcare resource consumption (outpatient and emergency room consultations) in order to evaluate its cost-efficiency compared to current standard interventions.

The study will include stable bipolar patients (YMRS ≤ 8, HDRS ≤ 6 for at least one month prior to study entry) who have experienced at least one hypomanic, manic or depressive relapse during the 12 months prior to study entry. This will be carried out in three different but complementary phases in order to fully include patients and therapist's preferences. Along the process, confidential information and data handling will be tested to ensure privacy and confidentiality are warranted. In this regard, an anonymized user name and password will be given to the patients who will never have to reveal their real identity to access the application during the study.

* First phase: During the first three months a feasibility study will be conducted evaluating the use, reliability and satisfaction monitoring symptoms (subjective information) using a smart-phone with the SIMPLe 1.0 application installed. The intervention will be consecutively offered to 30 stable adults (>18 years) fulfilling inclusion criteria. The patient will have to read and agree with the terms and sign an informed consent in order to participate. Sociodemographic data and standardized clinical as well as functional assessments will be administered at baseline, at the first, second and third month of the study. The assessments will include present manic symptoms using the Young Mania Rating Scale (YMRS), depressive symptoms using the Hamilton depression Rating Scale (HDRS), biological rhythms using the biological rhythms interview of assessment in neuropsychiatry (BRIAN), quality of life measured by World Health Organization quality of life assessment (WHOQOL-BREF) and treatment adherence using the Medication Adherence Rating Scale (MARS). A smart-phone device with the SIMPLe 1.0 application pre-installed, will be given to the participants for free during the study with the mandatory condition that it has to be their main mobile-phone during the next 3 months. In the case the patient accepts to participate but doesn´t want to switch from his/her current smart-phone, he/she will be offered the possibility to download the SIMPLe 1.0 application from the App Store and a username and password will be given to use it. The SIMPLe 1.0 application will ask the user by customizable automatic reminder notifications to answer daily and weekly questionnaires based on DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th edition) criteria for a manic, hypomanic, mixed or depressive episode. The use frequency will be measured by the daily and weekly questionnaires answered which will be registered online. At the same time they will receive through the application daily customized psychoeducative messages based on the information collected by the application. Feasibility and satisfaction will be assessed with the application usage log data and an electronic survey, while the app reliability to correctly asses the patients mood states will be analyzed comparing the clinical assessments and the information collected by the application.
* Second phase: Individual personal interviews with each SIMPLe 1.0 user will also collect qualitative information about the application and suggestions. Taking into consideration the information collected from participants in the first phase, the application will be adapted and improved with the addition of objective information (signs) monitoring modules using mobile usage parameters and the built-in sensors. Focus groups will be held with participants, psychiatrists and psychologists to better fit their needs and incorporate suggestions.
* Third phase: A randomized controlled trial taking into consideration a significance level of 0.05, power of 0.8 and a minimal detectable difference of 0.5 and an expected drop-out of 15%, will be carried out with two arms of 74 patients each, as follows:

  * Intervention group (SIMPLe 2.0 + TAU): The experimental group will use the application SIMPLe 2.0 and simultaneously will receive their usual treatment which includes pharmacological and psychological interventions. A smart-phone device with the SIMPLe 2.0 application pre-installed, will be given to the participants for free during the study with the mandatory condition that it has to be their main mobile-phone during the next 3 months. In the case the patient accept to participate but don´t want to switch from their current smart-phone, they will be offered the possibility to download the SIMPLe 2.0 application from the App Store and a username and password will be given to use it. The patient will be asked by customizable automatic reminder notifications to answer daily and weekly questionnaires based on DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th edition) criteria for a manic, hypomanic or depressive episode. Additionally, the signs will be automatically recorded based on the smart-phone usage measured by the smart-phone screen on time, texts messages sent, telephone calls made and social networking apps activity, in addition to the physical activity monitored by the built-in actimeter. At the same time, they will receive through the application daily psychoeducative customized messages based on the data recollected by the application. Relapse risk will be fixed by means of a logarithm including both subjective and objective data. If the logarithm points at a moderate or high risk, the clinical team will be immediately contacted and the patient will be offered to call emergency services for assistance.
  * Treatment as usual group (TAU): The treatment as usual (TAU) only group will be followed-up with their usual treatment including pharmacological and psychological interventions.

An initial evaluation in both groups will be carried out recollecting sociodemographic data and using standardized clinical as well as functional assessments which will be administered again in three follow-up evaluations, at three, six and twelve months. The assessments will include present manic symptoms using the Young Mania Rating Scale (YMRS), depressive symptoms using the Hamilton depression Rating Scale (HDRS), functional impairment using the Functioning assessment short test (FAST), biological rhythms using the biological rhythms interview of assessment in neuropsychiatry (BRIAN), quality of life measured by World Health Organization quality of life assessment (WHOQOL-BREF) and treatment adherence using the Medication Adherence Rating Scale (MARS). During the follow-up the number of relapses, inpatient admissions, outpatient consultations, emergency rooms consultations and suicide attempts will be registered. All participants in both groups must read and agree with the terms and sign an informed consent prior to their inclusion in the study. Psychiatrists and psychologists conducting the evaluations will be blinded to which participant belongs to each group.

The main outcome to evaluate between both groups during this period will be number of relapses (Manic, Hypomanic or Depressive Episodes) during the 6-month treatment phase. Secondary outcomes will include the number of relapses during 6-month post-intervention follow-up (Manic, hypomanic and depressive episodes according to DSM-5 criteria). In addition differences in biological rhythms (BRIAN), differences in manic symptoms using the Young Mania Rating Scale (YMRS) and depressive symptoms using the Hamilton depression Rating Scale (HDRS) during the 6-month treatment phase and 6-month post-intervention follow-up. Additionally the quality of life (WHOQOL-BREF), functional Impairment (FAST) and treatment adherence (Medication Adherence Rating Scale (MARS)) will be assessed each follow-up assessment. Other outcomes include differences in healthcare resource consumption measured in number and duration of hospitalizations, outpatient and emergency room consultations related to their psychiatric disorder and pharmacological treatment changes (doses and agents prescribed) over the 12 month follow-up.

In the case of positive results, the tested app will allow a user-friendly, non-costly and efficacious way to monitor and train stable bipolar patients avoiding recurrences, as an add-on to usual pharmacological care. The implementation of this technology will also improve associated healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the current diagnosis of Bipolar disorder type I or type II according to current DSM-5 criteria and confirmed with a semi structured interview (SCID).
* Hamilton Depression Scale score under or equal to 8 during the last month.
* Young Mania Rating Scale score under or equal to 6 during the last month.
* No history of relapses during the last 3 previous months but at least 1 relapse during the last year.
* Availability of a telephone account with an unlimited data plan during the 12 following months.

Exclusion Criteria:

* Lack of skills to use the offered smart-phone or unwillingness to learn them.
* FAST score above or equal to 20.
* Past or current participation in psychoeducation groups.
* Obsessive-compulsive disorder according to DSM-5 criteria.
* Concomitant severe medical condition.
* Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Estimated)
Dates: Start 2014-10; Primary Completion 2020-03 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Number of relapses during intervention | During the entire 6 months study period
  Number of relapses during intervention (manic, hypomanic and depressive episodes according to DSM-5 criteria).

SECONDARY OUTCOMES:
Biological rhythms | During the entire 6 months study period of the clinical trial and during 6-month post-intervention follow-up
  Difference in biological rhythms using the Biological Rhythms Interview of Assessment in Neuropsychiatry (BRIAN) during the entire 6 months study period of the clinical trial and during 6-month post-intervention follow-up.
Number of Relapses during 6-month post-intervention | 6-months post-intervention
  Number of Relapses during 6-month post-intervention follow-up (Manic, hypomanic and depressive episodes according to DSM-5 criteria).
Number of Manic and depressive symptoms | During the entire 6 months study period
  Difference in manic symptoms using the Young Mania Rating Scale (YMRS), depressive symptoms using the Hamilton depression Rating Scale (HDRS) during the entire 6 months study period.
Quality of life | During the entire 6 months study period of the clinical trial and during 6-month post-intervention follow-up
  Difference in quality of life measured by World Health Organization quality of life assessment (WHOQOL-BREF) during the entire 6 months study period of the clinical trial and during 6-month post-intervention follow-up.
Treatment adherence | During the entire 6 months study period of the clinical trial and during 6-month post-intervention follow-up
  Difference in treatment adherence using the Medication Adherence Rating Scale (MARS) during the entire 6 months study period of the clinical trial and during 6-month post-intervention follow-up.
Functional impairment | During the entire 6 months study period of the clinical trial and during 6-month post-intervention follow-up.
  Difference in functional impairment using the Functioning Assessment Short Test (FAST) during the entire 6 months study period of the clinical trial and during 6-month post-intervention follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Francesc Colom, PhD, Study Director — Institut Hospital del Mar d'Investigacions Mèdiques (IMIM); Eduard Vieta, MD, PhD, Study Chair — Hospital Clínic of Barcelona
Locations (1):
- Instituto Hospital del Mar de Investigaciones Médicas, Barcelona, Catalonia, Spain

REFERENCES:
- [Derived] Hidalgo-Mazzei D, Reinares M, Mateu A, Juruena MF, Young AH, Perez-Sola V, Vieta E, Colom F. Is a SIMPLe smartphone application capable of improving biological rhythms in bipolar disorder? J Affect Disord. 2017 Dec 1;223:10-16. doi: 10.1016/j.jad.2017.07.028. Epub 2017 Jul 10. PMID 28711743
- [Derived] Hidalgo-Mazzei D, Mateu A, Reinares M, Murru A, Del Mar Bonnin C, Varo C, Valenti M, Undurraga J, Strejilevich S, Sanchez-Moreno J, Vieta E, Colom F. Psychoeducation in bipolar disorder with a SIMPLe smartphone application: Feasibility, acceptability and satisfaction. J Affect Disord. 2016 Aug;200:58-66. doi: 10.1016/j.jad.2016.04.042. Epub 2016 Apr 20. PMID 27128358
- [Derived] Hidalgo-Mazzei D, Mateu A, Reinares M, Undurraga J, Bonnin Cdel M, Sanchez-Moreno J, Vieta E, Colom F. Self-monitoring and psychoeducation in bipolar patients with a smart-phone application (SIMPLe) project: design, development and studies protocols. BMC Psychiatry. 2015 Mar 20;15:52. doi: 10.1186/s12888-015-0437-6. PMID 25884824